CLINICAL TRIAL: NCT03280420
Title: Early Versus Late Catheter Removal in Patients With Acute Urinary Retention Secondary to Benign Prostatic Hyperplasia Under Tamsulosin Treatment
Brief Title: Early Versus Late Catheter Removal in Patients With Acute Urinary Retention Secondary to BPH Under Tamsulosin Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salem Hassan Salem Mohamed (Other)
Responsible Party: Sponsor-Investigator, Salem Hassan Salem Mohamed, Cairo, Egypt, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123urology
Record Dates: First submitted 2017-08-12; First posted 2017-09-12 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: BPH With Urinary Obstruction
Keywords: Acute urinary retention; BPH; TWOC; Tamsulosin

STUDY DESIGN:
Intervention Model Description: All patients were catheterized and received urinary antiseptic and then randomly divided into two groups : Group I :30 patients received Tamsulosin 0.4 mg once daily and catheter removed after 3 days. Group II :30 patients received Tamsulosin 0.4 mg once daily and catheter removed after 7 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early catheter removal (Active Comparator): 30 patients will receive Tamsulosin hydrochloride 0.4 mg once daily and the catheter will be removed after 3 days.
  Interventions: Procedure: Early catheter removal
- late catheter removal (Active Comparator): 30 patients will receive Tamsulosin hydrochloride 0.4 mg once daily and the catheter will be removed after 7 days.
  Interventions: Procedure: Late catheter removal

INTERVENTIONS:
Procedure: Early catheter removal — Patients will receive selective alpha blocker ( tamsulosin 0.4mg ) once daily and the catheter will be removed after 3 days.
  After catheter removal, patients will be allowed to void and will be discharged home who will have a successful void more than 200 cc of urine. Patients who will fail to void will be re-catheterized and will be prepared for prostatectomy.
  Other Names: After 3 days catheter removal
  Arms: early catheter removal
Procedure: Late catheter removal — Patients will receive selective alpha blocker ( tamsulosin 0.4mg ) once daily and the catheter will be removed after 7 days.
  After catheter removal, patients will be allowed to void and will be discharged home who will have a successful void more than 200 cc of urine. Patients who will fail to void will be re-catheterized and will be prepared for prostatectomy.
  Other Names: After 7 days catheter removal
  Arms: late catheter removal

SUMMARY:
The aim of this work is to compare between early (3days) and late(7days) removal of urinary catheter after acute urine retention in patients with Benign Prostatic Hyperplasia under Tamsulosin treatment.

DETAILED DESCRIPTION:
This is a prospective randomized study, Men with acute urinary retention secondary to benign prostatic hyperplasia were catheterized and then, if they fulfilled the entry criteria, were randomly assigned to receive 0.4 mg tamsulosin hydrochloride for three days or seven days, After that the catheter was removed and the ability to void unaided assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients having first attack of acute urinary retention secondary to BPH.

Exclusion Criteria:

* Renal impairment.
* Suspected urethral stricture.
* Neurogenic bladder.
* Cancer prostate.
* Medically induced retention.
* Previous use of alpha blockers.
* History of drug hypersensitivity or allergy to Tamsulosin.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-03-12 (Actual); Primary Completion 2017-09-16 (Actual); Study Completion 2017-09-16 (Actual)

PRIMARY OUTCOMES:
The duration for trial without catheter | 6 Months
  To determine the optimum period to remove catheter in patients complaining of acute urinary retention with benign prostatic hyperplasia.

SECONDARY OUTCOMES:
Factor affecting trial without catheter | 6 Months
  To evaluate the role of the following in trial without catheter patient's age prostate size residual urine volume prostatic specific antigen (PSA)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Badr, PHD, Study Chair — Al-Azhar University; Mohamed F El Saeed El Ebiary, MD, Study Director — Al-Azhar University
Locations (1):
- Faculty of medicine ,Al Azhar university, Cairo, El Mokhayam El Daem St.، Ezbet El-Arab, Nasr City, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT03280420/Prot_SAP_001.pdf